CLINICAL TRIAL: NCT02159612
Title: Disease Progression in Facioscapulohumeral Muscular Dystrophy - 1 Year MRI Follow-up
Brief Title: 1 Year MRI Followup in Facioscapulohumeral Muscular Dystrophy
Acronym: FSHD
Status: Completed | Type: Observational
Sponsor: Grete Andersen, MD (Other)
Responsible Party: Sponsor-Investigator, Grete Andersen, MD, Medical doctor, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Other Study IDs: H-3-2012-163 (fsh)
Record Dates: First submitted 2014-06-06; First posted 2014-06-10 (Estimated); Last update posted 2015-05-14 (Estimated); Status verified 2015-05

CONDITIONS: FSHD - Facioscapulohumeral Muscular Dystrophy
Keywords: FSHD; MRI; Disease progression
MeSH Terms: conditions — Muscular Dystrophy, Facioscapulohumeral; Disease Progression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- FSHD: A cohort of adult danish patients with facioscapulohumeral muscular dystrophy is invited to perform a MRI scan.
  Interventions: Other: MRI

INTERVENTIONS:
Other: MRI — MRI scan of muscles in the back and legs. Including T1, DIXON and STIR images.

SUMMARY:
An investigation of disease progression in adult danish patients with facioscapulohumeral muscular dystrophy. The disease progression is followed for a year with two test-days, including functional muscle tests and a MRI scan of muscles in the back and legs.

DETAILED DESCRIPTION:
A cohort of adult danish patients with facioscapulohumeral muscular dystrophy is invited to perform a MRI scan to describe the relation between backpain and disease affection in back muscles. After one year they are re-invited to perform another MRI scan to follow the disease progression.

The MRI scan is done to measure the quantity and quality of the muscles in the back, thigh and calf. Further, investigators investigate the muscle function by measuring of muscle strength in legs and in the back together with three functional tests. A walking test (6MWT), a stair test (14SST), and a chair test (5-TSTST). Self-assessment of back pain is measured by a standardized questionnaire about backpain.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with FSHD type 1

Exclusion Criteria:

* Pregnant or breastfeeding women.
* Patients with claustrophobia.
* Patients with implanted metallic parts in the body.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Persons in Denmark diagnosed with Facioscapulohumeral muscular dystrophy is invited to the study.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2014-05; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Fat infiltration | 1 year
  Change in the distribution of fat infiltration in back, thigh and calves muscles seen at the MRI images.

SECONDARY OUTCOMES:
Muscle structure | 1 year
  Muscle structure is evaluated with a four-point semi-quantitative visual scale. Two observers evaluate images independently. Changes in evaluation between 1st and 2nd scan are the outcome measure.
Muscle strength | 1 year
  Changes in muscle strength between 1st. and 2nd MRI-scan.
Back pain | 1 year
  Changes in self-assessed back-pain between 1st. and 2nd scan.
Muscle function | 1 year
  Changes in muscle function between 1st and 2nd MRI-scan, measured by a 6 minute walk test, a 14-step-stair test and a 5-times-sit-to-stand-test.

CONTACTS AND LOCATIONS:
Locations (1):
- Neuromuscular Research Unit, Department of Neurology, Rigshospitalet, Copenhagen, Denmark

REFERENCES:
- [Derived] Dahlqvist JR, Poulsen NS, Ostergaard ST, Fornander F, de Stricker Borch J, Danielsen ER, Thomsen C, Vissing J. Evaluation of inflammatory lesions over 2 years in facioscapulohumeral muscular dystrophy. Neurology. 2020 Sep 1;95(9):e1211-e1221. doi: 10.1212/WNL.0000000000010155. Epub 2020 Jul 1. PMID 32611642
- See also: The home-page of neuromuscular research units department in Copenhagen, Denmark — http://neuromuscular.dk